CLINICAL TRIAL: NCT06105346
Title: Prevalence Study of ENT-related Diseases in Conscripts at the Military Induction Board
Brief Title: Prevalence of ENT Diseseas
Acronym: PrENT
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: PrENT v1
Record Dates: First submitted 2023-10-09; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Conscripts; Military Induction Board; ENT Disease; Rhinosinusitis Chronic; Rhinosinusitis; HPV Infection; HPV Vaccine; Long COVID; ENT Surgery
Keywords: ENT; prevalence; military induction board; conscripts; rhinosinusitis; Long COVID; ENT surgeries; HPV vaccination; inborn hearing loss
MeSH Terms: conditions — Otorhinolaryngologic Diseases; Rhinosinusitis; Papillomavirus Infections; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study will be to evaluate in conscripts at the military induction board the prevalence of rhinosinusitis, the prevalence of HPV vaccinations, the prevalence of hearing impairments and the prevalence of long-COVID symptoms and further, to evaluate different factors that influence on the one hand the prevalence (urban-bred, non-urban-bred) and on the other hand symptoms (ENT-surgeries in medical history). Further, we want to evaluate if there is a correlation between subjective symptoms and apparated-based diagnostic investigations.

Therefore, questionnaires and data of medical examinations, aquired routinely at the military induction board, will be analysed.

DETAILED DESCRIPTION:
Rhinosinusitis is a very common complaint at ENT departments, whereby symptoms of the underlying disease are varying. Therefore, there is growing interest in prevalence of rhinosinusitis including differences in prevalence's depending on where the patient grew up. Further, there is growing interest in answering the question if different factors, including ENT-surgeries in medical history have an impact on symptoms of rhinosinusitis.

Within the past few years there is growing interest in carring out as many HPV-vaccinations as possible in order to reduce the prevalence of HPV-associated cancers.

Further, in adolescents there is a growing number of hearing impairments, including hearing loss and/or sounds in the ears.

Next, since the beginning of the COVID pandemic there are very common complaints in adult and pediatric patients about persistent medical problems for weeks or months after an acute SARS-CoV-2-infection and cannot be explained by another diagnosis, called long- Covid disease.

The military induction board of conscripts enables access to data from a cross-section of the population, with common characteristics of gender and age.

In the present study we want therefore to evaluate in conscripts at the military induction board the prevalence of rhinosinusitis, the prevalence of HPV vaccinations, the prevalence of hearing impairments and the prevalence of long-COVID symptoms and further, to evaluate different factors that influence on the one hand the prevalence (urban-bred, non-urban-bred) and on the other hand symptoms (ENT-surgeries in medical history). Further, we want to evaluate if there is a correlation between subjective symptoms and apparated-based diagnostic investigations.

ELIGIBILITY:
Inclusion Criteria:

* participation of the military induction board of conscripts
* consent for participation obtained by the conscripts
* completed questionnaire (with at least 50% completeness of each subcategory)
* participation of medical examination

Exclusion Criteria:

* no consent for participation in the study by the conscripts
* incomplete questionnaire (with less than 50% completeness of each subcategory)
* no participation of medical examination.

Ages: 17 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — only Austrian males (conscripts), who are invited at the military induction board
Study Population: All male Austrian conscripts who take part at the military inductions board are eligible for the study inclusion.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of rhinosinusitis | Through data collection, an average of 1 week
  To assess whether there is a difference in prevalence of rhinosinusitis in urban-bred conscripts compared to non-urban-bred conscripts.
Prevalence of human papilloma virus vaccination | Through data collection, an average of 1 week
  To assess whether there is a difference in prevalence of human papilloma virus vaccinations in urban-bred conscripts compared to non-urban-bred conscripts.
Prevalence of hearing impairment | Through data collection, an average of 1 week
  To assess whether there is a difference in prevalence of hearing impairment in urban-bred conscripts compared to non-urban-bred conscripts.
Prevalence of long-COVID disease | Through data collection, an average of 1 week
  To assess whether there is a difference in prevalence of long-COVID disease in vaccinated conscripts compared to no-vaccinated conscripts.

SECONDARY OUTCOMES:
Prevalence of rhinosinusitis | Through data collection, an average of 1 week
  To assess prevalence of rhinosinusitis in conscripts at the military induction board
Prevalence of rhinosinusitis | Through data collection, an average of 1 week
  To assess the different symptoms of rhinosinusitis in conscripts at the military induction board
Prevalence of rhinosinusitis | Through data collection, an average of 1 week
  To assess the prevalence of rhinosinusitis in conscripts with previous ENT-surgeries
Prevalence of rhinosinusitis | Through data collection, an average of 1 week
  To assess differences in symptoms in rhinosinusitis in conscripts with previous ENT-surgeries
Prevalence of rhinosinusitis | Through data collection, an average of 1 week
  To assess the combined prevalence of rhinosinusitis and chronic pulmonary diseases in conscripts
Prevalence of rhinosinusitis | Through data collection, an average of 1 week
  To assess the difference in prevalence of subjective symptoms of rhinosinusitis compared to objective (apparatus based and laboratory based) symptoms of rhinosinusitis
Prevalence of rhinosinusitis | Through data collection, an average of 1 week
  To analyse demographic data in conscripts with rhinosinusitis
Prevalence of human papilloma virus vaccines | Through data collection, an average of 1 week
  To assess the prevalence of HPV vaccines among conscripts at the military induction board
Prevalence of human papilloma virus vaccines | Through data collection, an average of 1 week
  To assess knowledge about HPV and HPV vaccinations and in dependent of that prevalence of HPV vaccines among conscripts at the military induction board
Prevalence of hearing impairment | Through data collection, an average of 1 week
  To assess the prevalence of hearing impairment in conscripts at the military induction board
Prevalence of hearing impairment | Through data collection, an average of 1 week
  To assess the difference in prevalence of subjective symptoms of hearing impairment compared to objective (apparatus based and laboratory based) signs of hearing impairment
Prevalence of hearing impairment | Through data collection, an average of 1 week
  To analyse demographic data in conscripts with hearing impairment
Prevalence of long-COVID | Through data collection, an average of 1 week
  To assess the prevalence of long-COVID in conscripts at the military induction board
Prevalence of long-COVID | Through data collection, an average of 1 week
  To assess different symptoms of long-COVID in conscripts at the military induction board
Prevalence of COVID-19 infection | Through data collection, an average of 1 week
  To assess the prevalence of previous COVID 19 infections in conscripts at the military induction board
Prevalence of long-COVID | Through data collection, an average of 1 week
  To analyse demographic data in conscripts with long-COVID